CLINICAL TRIAL: NCT06255340
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 3031185 Administered as Tablet to Healthy Male Subjects, and a Randomised, Open-label, Single-dose, Two-way Cross-over Relative Bioavailability Comparison of BI 3031185 as Tablet With and Without Food in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 3031185 Are Tolerated and How Food Influences the Amount of BI 3031185 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1516-0001
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The food effect (FE) part of the trial is designed as a randomised, two-sequence, open-label, two period, two-way cross-over trial.
  The single rising dose (SRD) part is designed as blinded to subjects, randomised, and placebo-controlled within parallel dose groups.
Masking Description: FE part of the trial is designed as open-label. SRD part is designed as blinded to subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- SRD Part: BI 3031185 dose group 1 (Experimental): Single rising dose (SRD)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 2 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 3 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 4 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 5 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 6 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 7 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: BI 3031185 dose group 8 (Experimental)
  Interventions: Drug: BI 3031185
- SRD Part: Placebo matching BI 3031185 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3031185
- FE part: BI 3031185 under fasted (Reference, R) then BI 3031185 under fed (Test,T) conditions (Experimental): Food effect (FE)
  Interventions: Drug: BI 3031185
- FE part: BI 3031185 under fed (Test,T) then BI 3031185 under fasted (Reference, R) conditions (Experimental)
  Interventions: Drug: BI 3031185

INTERVENTIONS:
Drug: BI 3031185 — BI 3031185
  Arms: FE part: BI 3031185 under fasted (Reference, R) then BI 3031185 under fed (Test,T) conditions; FE part: BI 3031185 under fed (Test,T) then BI 3031185 under fasted (Reference, R) conditions; SRD Part: BI 3031185 dose group 1; SRD Part: BI 3031185 dose group 2; SRD Part: BI 3031185 dose group 3; SRD Part: BI 3031185 dose group 4; SRD Part: BI 3031185 dose group 5; SRD Part: BI 3031185 dose group 6; SRD Part: BI 3031185 dose group 7; SRD Part: BI 3031185 dose group 8
Drug: Placebo matching BI 3031185 — Placebo
  Arms: SRD Part: Placebo matching BI 3031185

SUMMARY:
This trial starts the clinical development of BI 3031185. The single rising dose (SRD) part of the trial investigates safety, tolerability, and pharmacokinetics of a range of single doses of BI 3031185 as basis for further development.

The food effect (FE) part is conducted to assess the effect of food on the relative bioavailability of the BI 3031185 tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests without any clinically significant abnormalities
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 89 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease. This does not include acceptable concomitant conditions that were not assessed as clinically relevant by the investigator (e.g. possible cases of myopia, hyperopia, astigmatism, non-active pollinosis, or mild acne of the skin)
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
SRD part: The occurrence of any treatment-emergent adverse event (AE) assessed as drug-related by the investigator | Up to 22 days
FE part: Area under the concentration-time curve of the analyte in plasma over the dosing interval 0 to 24 hours (AUC0-24) | Up to 24 hours
FE part: Maximum measured concentration of the analyte in plasma (Cmax) | Up to 8 days

SECONDARY OUTCOMES:
SRD part: Area under the concentration-time curve of the analyte in plasma over the dosing interval 0 to 24 hours (AUC0-24) | Up to 24 hours
SRD part: Maximum measured concentration of the analyte in plasma (Cmax) | Up to 13 days
FE part: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com